CLINICAL TRIAL: NCT00376610
Title: Prospective Clinical Evaluation of ASR/Re-Cap Resurfacing Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KF1127957
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2007-07-04 (Estimated); Status verified 2007-07

CONDITIONS: Bearings

INTERVENTIONS:
Device: ASR/Re-cap

SUMMARY:
ASR/Re-cap versus 28 MoM

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of THA
* ASA I-II
* Willing to return for follow-up evaluations

Exclusion Criteria:

* Collum femurs < 2 cm
* Cysts > 1 cm
* Caput necrose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Arne Borgwardt, Study Director — Frederiksberg Univesity Hospital
Locations (1):
- Frederiksberg University Hospital, Frederiksberg, Copenhagen, Denmark